CLINICAL TRIAL: NCT06374472
Title: Surgical Treatment of Fractures of the Dorso-lombar Spine
Status: Completed | Type: Observational
Sponsor: Ibn Jazzar Hospital (Other)
Responsible Party: Principal Investigator, Zied Mansi, Principal investigator, Ibn Jazzar Hospital
Other Study IDs: IRB00001194
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Spine Fracture
Keywords: Fractures; Spine; Surgery; Treatment; Evaluation; Results
MeSH Terms: conditions — Spinal Fractures; Fractures, Bone | interventions — Fracture Fixation, Internal; Arthrodesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 80 cases of thoracolumbar spine fractures
  Interventions: Procedure: Osteosynthesis

INTERVENTIONS:
Procedure: Osteosynthesis — Some patients had osteosynthesis using a long construct, others had osteosynthesis using a short construct. Short constructs designated constructs only taking one level above and one level below the injury level (the fractured vertebra was not always included in the construct). The montages taking more than one level above or below the lesion were considered to be a long montage. Osteosynthesis is carried out using Cotrel Dubousset type rods and screws.
  Other Names: Release gestures; Arthrodesis; First approach

SUMMARY:
Trauma to the thoracolumbar spine is responsible for potentially serious lesions, most often involving the functional prognosis in the short, medium and long term, and rare The frequency of these traumas is explained by falls from high places, especially during work accidents or suicide attempts, but also by the perpetual increase in accidents on public roads ly the vital prognosis

DETAILED DESCRIPTION:
Trauma to the thoracolumbar spine is responsible for potentially serious lesions, most often involving the functional prognosis in the short, medium and long term, and rarely the vital prognosis .

The thoracolumbar spine has an extended transition zone between the tenth thoracic vertebra (T10) and the second lumbar vertebra (L2): the thoracolumbar hinge which, given its particular anatomical situation between a poorly mobile thoracic segment and a dynamic lumbar segment, is the predilection for occurrence of fractures and dislocations .

The frequency of these traumas is explained by falls from high places, especially during work accidents or suicide attempts, but also by the perpetual increase in accidents on public roads.

The analysis of the lesion mechanism and its consequences depends on the understanding of the classification of these lesions which are essential for therapeutic conduct .

Surgical treatment constitutes a key element in the management strategy for these fractures

ELIGIBILITY:
Inclusion Criteria:

* the files of patients hospitalized for a recent fracture of the thoracolumbar spine within 12 months

Exclusion Criteria:

* Files with insufficient follow-up, patients lost to follow-up. patients presenting: A pathological fracture. Osteoporotic collapse. Material and Methods 3 Staged trauma to the spine. A fracture due to ankylosing spondylitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 80 cases of surgically treated thoracolumbar spine fractures
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Age (in years) | from enrollment to the end of treatment at 4 years
  average age of our patients was 38.25 years with extremes of 16 years and 68 years
Sex | from enrollment to the end of treatment at 4 years
  Our series is characterized by a significant male predominance, it included 47 men (58.75%) and 33 women (41.25%), with a sex ratio of 1.42
Neurological status ( Frenkel classification) | from enrollment to the end of treatment at 4 years
  3 Frankel A patients, 1 Frankel B patient, 6 Frankel C patients and 6 Frankel D

CONTACTS AND LOCATIONS:
Locations (1):
- IBN jazzar hospital, Kairouan, Tunisia

IPD SHARING:
Plan to Share IPD: No
further use of this informations for others group works